CLINICAL TRIAL: NCT05976503
Title: A Randomized, Blind, Placebo-controlled, Three-way Crossover Study to Evaluate the Potential Interaction of Tunodafil Hydrochloride Tablets and Alcohol in Healthy Chinese Male Participants
Brief Title: A Study of the Interaction of Tunodafil Hydrochloride Tablets and Alcohol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YZJ-YKNF-DDI-08
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tunodafil Hydrochloride plus alcohol (Experimental): Participants received 100 mg Tunodafil Hydrochloride Tablets plus 0.5 g/kg alcohol.
  Interventions: Drug: Tunodafil Hydrochloride Tablets; Other: Alcohol
- Placebo plus alcohol (Experimental): Participants received placebo plus 0.5 g/kg alcohol.
  Interventions: Drug: Placebo; Other: Alcohol
- Tunodafil Hydrochloride (Experimental): Participants received 100mg Tunodafil Hydrochloride Tablets.
  Interventions: Drug: Tunodafil Hydrochloride Tablets

INTERVENTIONS:
Drug: Tunodafil Hydrochloride Tablets — 100mg Tunodafil Hydrochloride Tablets
  Arms: Tunodafil Hydrochloride; Tunodafil Hydrochloride plus alcohol
Drug: Placebo — Placebo
  Arms: Placebo plus alcohol
Other: Alcohol — 0.5 g/kg alcohol
  Arms: Placebo plus alcohol; Tunodafil Hydrochloride plus alcohol

SUMMARY:
The purpose of this study is primarily to evaluate the effects of simultaneous administration of Tunodafil Hydrochloride Tablets with alcohol on blood pressure, pulse rate and pharmacokinetics in healthy Chinese male participants.

DETAILED DESCRIPTION:
This study will be divided into two parts: pre-trial and formal trial. The pre-trial is a non-randomized, open design to evaluate the safety and tolerability of Tunodafil Hydrochloride Tablets in combination with alcohol in healthy male participants. Four participants will be taken 50mg or 100mg doses with alcohol. Supine blood pressure (systolic and diastolic), pulse rate, PK blood sample collection should be performed before and after administration, and the time point is the same as the formal trial.

The dosage of Tunodafil Hydrochloride Tablets in the formal trial will be determined based on the pre-trial results.

The formal trial is a single-center, randomized, blind, placebo-controlled, three-cycle crossover design, and 18 participants will be randomized to receive the following three treatments. The test is administered once per cycle and the washout period is 7 days:

Treatment A: A single oral dose of Tunodafil Hydrochloride Tablets plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).

Treatment B: A single oral dose of placebo plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).

Treatment C: A single oral dose of Tunodafil Hydrochloride Tablets plus an oral dose of placebo drink mixed with fruit juice.

For each treatment period, supine blood pressure and pulse rate will be measured at pre-dose and up to 24 hours post-dose. Blood will be collected at pre-dose and up to 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who can understand and are willing to strictly follow the clinical trial protocol to complete the trial and sign the informed consent;
2. Male participants aged 18~45 years (including the cut-off value);
3. Weight≥50.0kg; Body mass index (BMI) in the range of 19.0~26.0kg/m^2 (including the critical value);
4. Good health, no history of respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system and other serious diseases or chronic diseases;
5. Do not plan to have children during the trial, and agree to use reliable contraception during the trial and for 3 months after the last study drug administration, and do not plan to donate sperm.

Exclusion Criteria:

1. Allergic: allergic to drugs, food, pollen, alcohol, etc., known to be allergic to experimental drugs or other PDE5 inhibitors and excipients;
2. Patients with difficulty swallowing tablets/capsules; Or according to 0.5g/kg body weight intake of alcohol (that is, 70kg body weight participants drink 35g pure alcohol, equivalent to 50 degrees of liquor about 70g) may be intoxicated; Or have special dietary requirements and cannot accept the standard diet provided by the research center;
3. Patients who have a history of needle fainting and blood fainting, can not tolerate venous puncture blood collection and/or have difficulty in blood collection;
4. Patients with abnormal color vision judged by researchers to have clinical significance; Or have known to have retinitis pigmentosa, macular degeneration, nonarteriotic anterior ischemic optic neuropathy (NAION) eye disease; Or have known fundus medical history that other investigators have deemed unsuitable for inclusion;
5. People who have experienced sudden hearing loss or hearing loss in the past;
6. Past or existing postural hypotension/syncope;
7. Clinically significant vital signs (reference value range: 90 mmHg≤systolic blood pressure (sitting) <140 mmHg, 60 mmHg≤diastolic blood pressure (sitting)<90 mmHg, 55 times/min≤pulse rate (resting)≤100 times/min, 35.5℃≤body temperature (axillary temperature)≤37.2℃; Participant to the judgment of the study physician); Or physical examination, 12-lead electrocardiogram, laboratory test results, the investigator judged that the abnormality is clinically significant;
8. Hepatitis B virus surface antigen, hepatitis C virus antibody, treponema pallidum specific antibody, human immunodeficiency virus antibody any abnormal clinical significance;
9. Those who have used soft drugs (such as cannabis) within 3 months before screening or hard drugs (such as cocaine, amphetamines, Phencyclidine, etc.) within 1 year before screening; Or have a history of drug abuse; Or positive urine drug screening before randomization;
10. Positive breath test for alcohol;
11. Smokers who have smoked more than 5 cigarettes per day in the 3 months before screening or could not stop using any tobacco products during the test;
12. Participants in any clinical trial within 3 months prior to screening;
13. Those who have participated in blood donation and total blood donation or total blood loss≥400mL within 3 months before screening, or participated in blood donation and total blood donation≥200mL or total blood loss≥200mL within 1 month; Or receiving blood transfusion; Or plan to donate blood within 1 month after the end of this trial;
14. Those who have undergone surgery within 30 days prior to screening, or plan to undergo surgery during the trial;
15. Those who have received vaccination within 30 days prior to screening, or who plan to receive vaccination during the trial;
16. Use of any CYP3A4/5 inhibitors or inducers (e.g., inhibitors-itraconazole, fluconazole, clarithromycin, ritonavir, cimetidine, diltiazem, etc.) within 28 days prior to randomization; Inducers-rifampicin, phenobarbital, carbamazepine);
17. Those who have taken any prescription drugs, non-prescription drugs, health products, vitamins, or Chinese herbs within 14 days before randomization;
18. Those who have eaten grapefruit, pomelo, dragon fruit, mango and other fruits or related products that affect metabolic enzymes within 7 days before randomization;
19. People who ingested beverages or foods rich in caffeine or xanthine (such as coffee, strong tea, chocolate, cola, etc.) within 48 hours before randomization;
20. Patients who developed acute disease from the screening stage to before randomization;
21. Participants judged by the investigator to be unsuitable for this clinical trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sexes Eligible for the Study
Enrollment: 22 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Maximum change in systolic blood pressure (SBP) | 4 hours after treatment
  Maximum change from baseline in decubitus (semi-decubitus) SBP.
Maximum change in diastolic blood pressure (DBP) | 4 hours after treatment
  Maximum change from baseline in decubitus (semi-decubitus) DBP.
Maximum change in pulse | 4 hours after treatment
  Maximum change from baseline in decubitus (semi-decubitus) position.
The area under effect-time curve (AUEC0- 4h) of supine SBP | 4 hours after treatment
  The area under effect-time curve (AUEC0- 4h) of supine SBP relative to baseline change.
The area under effect-time curve (AUEC0- 4h) of supine DBP | 4 hours after treatment
  The area under effect-time curve (AUEC0- 4h) of supine DBP relative to baseline change.
The area under effect-time curve (AUEC0- 4h) of pulse | 4 hours after treatment
  The area under effect-time curve (AUEC0- 4h) of pulse relative to baseline change.
Peak concentration (Cmax) of Tunodafil and metabolites M459 | 24 hours after treatment
Area under drug time curve (AUC) of Tunodafil and metabolites M459 | 24 hours after treatment
Peak concentration (Cmax) of alcohol | 8 hours after treatment

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0 | 7 days after treatment
  A treatment-emergent adverse events (TEAE) is defined as any unfavorable and unintended sign,symptom or disease temporally associated with the use of a study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China